CLINICAL TRIAL: NCT06940245
Title: Motor and Cognitive Abilities in Relation to Fall Risk: Use of Virtual Reality for the Assessment of Attentional and Reaction Capacities
Brief Title: Use of Virtual Reality for the Assessment of Attentional and Reaction Abilities for Fall Risk Evaluation
Status: Not yet recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: VR&RISKofFALL
Record Dates: First submitted 2025-04-02; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Aging; Fall Risk Factors; Sleep

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Aging is a condition characterized by a general decline in physical and cognitive performance, however its effects on various functions are still controversial. These changes lead to an increased risk of injuries, particularly due to falls. According to the World Health Organization (WHO) report, 28-35% of individuals aged over 65 experience a fall each year, and this percentage increases with age. For this reason, preventing falls among the elderly is undeniably one of the most critical public health issues in today's aging society. Nowadays, it is widely demonstrated that the loss of muscle strength and mass, along with decreased balance, significantly increases the risk of falls. However, with aging, numerous other changes occur that contribute to an increased risk of falls, such as a decline in cognitive function, including attention, reaction capabilities and memory, as well as other factors that worsen the quality of life, such as insufficient sleep or nutrition. According to WHO estimates, by 2030, the number of injuries due to falls will double. Therefore, it is of great importance to understand and analyze the factors contributing to falls among older adults in everyday life. For this reason, the principal aim of this study was to evaluate the correlation between the fall index and the Visual Attention, Reaction Time and visual field using the technologies of Virtual Reality (VR). Since aging brigs changes in different aspect, the secondary objectives aim to study the correlation also with i) sleep quantity and quality parameters, ii) risk of malnutrition, and iii) physical condition, muscle conditions and strength in order to have a comprehensive understanding of the factors that most contribute to the risk of falls. In addition to these objectives, the correlation between acute sleep deprivation and the risk of falls will also be analyzed, in order to understand how inadequate sleep quantity can impact injuries in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any ethnicity;
* Age ≥ 60 years;
* Cognitively intact;
* Autonomous ambulation;
* Signed and accepted informed consent to participate in all procedures required for the study.

Exclusion Criteria:

* Body Mass Index > 40.0;
* History of epileptic episodes;
* Bone fractures in the last 6 months;
* Previous surgical treatments for orthopedic conditions performed in the six months prior to study inclusion;
* Use of medications that affect motor coordination, balance, and bone and muscle metabolism;
* Conditions that, despite autonomous ambulation, influence fall risk (e.g., orthopedic, rheumatologic, or neurological conditions);
* Carriers of pacemakers and mechanical implants.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 100 subjects aged 60 years or older will be recruited, but recruitment will continue until enough subjects are identified to reach the predetermined number for the second study. The subjects are chosen on the basis of the following inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
30 - second chair stand test | 10 days ± 3 days after the familiarization day
  to assess the leg strength and endurance in older adults. Being in a specific sitting position on a chair, the test consists of getting up and sitting down as many times as possible in 30 seconds

SECONDARY OUTCOMES:
Virtual reality (VR-Brain Tracker) | 10 days ± 3 days after the familiarization day
  Evaluation to assess visual attention through the Multiple Object Tracking paradigm.
Strength asessment | 10 days ± 3 days after the familiarization day
  Handgrip Test (Kg) Flexors and Extensors of thigh muscles (Kg)
Balance test | 10 days ± 3 days after the familiarization day
  balance assessment is conducted using Baiobit equipment from BTS Bioengineering. The maximal balance time in monopodalic will be considered (s)
Sleep assessment | sleep monitoring duration: 10 days ± 3 days after the familiarization day
  Objective assessment of sleep quantity and quality using the MotionWatch 8® (CamTec, USA), and sleep diary.
Sleep Hygene Index | 10 days ± 3 days after the familiarization day
  Questionnaire to assess the sleep hygene
Body Impedence Assessment | T1
  to assess body composition by measuring the resistance of electrical flow through the body. It helps estimate parameters like body fat percentage, muscle mass, and water content. BIA is commonly used in health and fitness settings to monitor changes in body composition, guide nutritional and fitness plans, and assess overall health.
Virtual reality (CNS Sprint) | 10 days ± 3 days after the familiarization day
  To assess the response time (ms)
Virtual reality (Visual efficiency) | 10 days ± 3 days after the familiarization day
  To assess the visual field
The Pittsburgh Sleep Quality Index | 10 days ± 3 days after the familiarization day
  Questionnaire to assess sleep quality
Morningness-Eveningness Questionnaire | 10 days ± 3 days after the familiarization day
  Questionnaire to assess the chronotype
Karolinska Sleepiness Scale | 10 days ± 3 days after the familiarization day
  Scale to assess the sleepiness
Tiredness Severity Scale | 10 days ± 3 days after the familiarization day
  Scale to assess the tiredness
SARC-F | 10 days ± 3 days after the familiarization day
  A QUESTIONNAIRE FOR SCREENING THE RISK OF SARCOPENIA
International Physical Activity Questionnaire | 10 days ± 3 days after the familiarization day
  Questionnaire to assess the physical activity
BORG-CR10 scale | 10 days ± 3 days after the familiarization day
  EFFORT PERCEPTION SCALE
Mini Nutritional Assessment | 10 days ± 3 days after the familiarization day
  QUESTIONNAIRE TO ASSESS THE RISK OF MALNUTRITION
Nutritional diary | 10 days ± 3 days after the familiarization day
  Keeping a food diary helps collect accurate data on participants' eating habits for scientific analysis.

IPD SHARING:
Plan to Share IPD: Undecided